CLINICAL TRIAL: NCT00594581
Title: A Single-Site, Double-Blind, Phase II Trial to Investigate the Safety, Toleration, Systemic Exposure and Anti-Scarring Potential of Different Applications of Intradermal Juvista (Avotermin) in Male Subjects Aged 18-45 Years
Brief Title: Anti-Scarring Efficacy and Safety of Intradermal Juvista (Avotermin) in Healthy Males
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Renovo (Industry)
Responsible Party: Mark Cooper, SVP of Clinical Operations, Renovo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RN1001-319-1011
Record Dates: First submitted 2007-12-11; First posted 2008-01-15 (Estimated); Last update posted 2008-01-15 (Estimated); Status verified 2008-01

CONDITIONS: Cicatrix
Keywords: cicatrix, scarring, TGF-beta3, avotermin, Juvista
MeSH Terms: conditions — Cicatrix; Arrhythmogenic Right Ventricular Dysplasia, Familial, 1 | interventions — TGFB3 protein, human; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Juvista (avotermin) 50ng/100μl/linear cm wound margin
  Interventions: Drug: Juvista (avotermin) plus placebo, standard-care (within-subject controls)
- 2 (Active Comparator): Juvista (avotermin) at 200ng/100μl/linear cm
  Interventions: Drug: Juvista (avotermin) plus placebo, standard-care (within-subject controls)

INTERVENTIONS:
Drug: Juvista (avotermin) plus placebo, standard-care (within-subject controls) — Intradermal Juvista (avotermin) at 50ng or 200ng per 100μl per linear cm of wound margin
  Other Names: Juvista; RN1001; Avotermin

SUMMARY:
This study was undertaken to investigate safety and scar-improvement activity of different applications of Juvista (avotermin), administered to surgical incisions made to the skin of a healthy population of male volunteers aged 18-45 years. The study addressed two issues: whether Juvista (avotermin) administered at 200ng/100μl/linear cm wound margin is more effective than 50ng/100μl/linear cm for scar improvement and, secondly, whether dosing once only (before wounding) or twice (before and after wounding) is optimal for scar improvement.

ELIGIBILITY:
Inclusion Criteria:

* Clinically healthy, male subjects aged 18 to 45 years (inclusive)
* Body weight between 40kg and 150kg or a body mass index within the range 15-55kg/m2, calculated using Quetelet's index

Exclusion Criteria:

* Subjects with history or evidence of hypertrophic or keloid scarring, or with tattoos or previous scars in the area to be biopsied.
* Subjects with tattoos or previous scars within 3cm of the area to be incised during the trial.
* Afro-Caribbean volunteers, because of their increased susceptibility to hypertrophic and keloid scarring.
* Subjects who, on direct questioning and physical examination, have evidence of any past or present clinically significant disease.
* Subjects with a chronic or currently active skin disorder, which would adversely affect the healing of the acute wounds or involved the areas to be examined in this trial.
* Subjects with a history of clinically significant allergies.
* Subjects with any clinically significant abnormality following review of pre-trial laboratory data and physical examination.
* Subjects taking, or who had taken, certain prescribed drugs in the 4 weeks before to Day 0 and, in particular, topical or systemic steroids, anti-inflammatory, anti-coagulant, anti-proliferative drugs, and antibiotics.
* Subjects who have taken part in a clinical trial within 3 months before admission to this trial, or who are currently participating in a clinical trial, whether an investigational drug was involved or not.
* Subjects with any clinical evidence of severe ongoing, or prolonged, depression or mental illness.
* Subjects smoking more than 20 cigarettes a day.
* Subjects drinking more than 28 units of alcohol per week (1 unit = ½ pint of beer [285ml], 25ml of spirits, or 1 glass of wine).
* Subjects showing evidence of drug abuse.
* Subjects known to have, or to have had, serum hepatitis or who were carriers of the hepatitis B surface antigen (HbsAg) or hepatitis C antibody.
* Subjects previously testing positive for HIV antibodies, or who admit to belonging to a high-risk group.
* Subjects with pre-existing clinically significant neurological conditions.
* Subjects who, in the opinion of an investigator, are not likely to complete the trial for whatever reason.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2003-10; Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Scar appearance | 12 months

SECONDARY OUTCOMES:
Safety: adverse events, local tolerability, systemic exposure | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jim Bush, MBChB, Principal Investigator — Renovo Ltd
Locations (1):
- Clinical Trials Unit, Renovo Ltd, Manchester, La, United Kingdom

REFERENCES:
- [Derived] Bush J, Duncan JAL, Bond JS, Durani P, So K, Mason T, O'Kane S, Ferguson MWJ. Scar-improving efficacy of avotermin administered into the wound margins of skin incisions as evaluated by a randomized, double-blind, placebo-controlled, phase II clinical trial. Plast Reconstr Surg. 2010 Nov;126(5):1604-1615. doi: 10.1097/PRS.0b013e3181ef8e66. PMID 21042116